CLINICAL TRIAL: NCT01490905
Title: A Double Blind Placebo Study to Determine the Effectiveness of Theramine on the Management of Chronic Back Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Targeted Medical Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0820102
Record Dates: First submitted 2011-11-22; First posted 2011-12-13 (Estimated); Last update posted 2011-12-13 (Estimated); Status verified 2011-12

CONDITIONS: Chronic Low Back Pain
Keywords: Medical food; Theramine; Ibuprofen; Amino acids; Convenience Pack Kit
MeSH Terms: interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Theramine active and ibuprofen placebo (Active Comparator): 2 capsules Theramine twice daily with one ibuprofen-like placebo once daily.
  Interventions: Other: Theramine (A medical food)
- Theramine and Ibuprofen (Theraprofen) (Active Comparator): Two capsules Theramine twice daily with Ibuprofen 400mg once daily.
  Interventions: Drug: Theraprofen
- Theramine placebo and Ibuprofen (Active Comparator): Two Theramine-like placebo twice daily and one ibuprofen 400mg.
  Interventions: Drug: Ibuprofen

INTERVENTIONS:
Other: Theramine (A medical food) — Theramine two capsules twice daily for 28 days.
  Arms: Theramine active and ibuprofen placebo
Drug: Theraprofen — Theramine two capsules twice daily and ibuprofen 400mg once daily for 28 days.
  Arms: Theramine and Ibuprofen (Theraprofen)
Drug: Ibuprofen — Ibuprofen 400mg once daily for 28 days.
  Arms: Theramine placebo and Ibuprofen

SUMMARY:
This research protocol will compare Theramine to a non-steroidal anti-inflammatory drug (NSAID) in the treatment of chronic back pain. The study will examine the efficacy and tolerability of Theramine alone in patients with chronic back pain in comparison to the NSAID, Ibuprofen, and the co-administration of Ibuprofen with Theramine.

DETAILED DESCRIPTION:
The diagnosis and management of back pain is a challenge for both primary care physicians and specialists. Establishing an etiology can be difficult and often problematic, with treatment options capable of producing serious and potentially life threatening side effects. Treatments often exert a modest impact on the natural history of the condition. Non-steroidal anti-inflammatory drugs (NSAIDs) are frequently prescribed to treat chronic back pain. NSAIDs are only moderately effective in relieving pain. NSAIDs are the leading cause of drug-induced gastrointestinal bleeds, the most common cause of drug-induced morbidity and mortality particularly at high dose. They can also exacerbate hypertension, edema and produce nephrotoxicity. The effects are also dose dependent. Recent data indicates NSAIDs are a risk factor for myocardial infarction, particularly at high doses. Recent data also indicates NSAIDs disrupt collagen repair in injured tissue. Muscle relaxants and narcotic analgesics show limited efficacy and often produce sedation, constipation or inappropriate usage. Physical therapy and local modalities often are not satisfying, costly, and require considerable investment of patient time.

Neurotransmitter depletion has been demonstrated to contribute to chronic pain states. Increased nutrient requirements associated with pain syndromes and the consequent reduced production of neurotransmitters contribute to maladaptive pain responses. The ability to enhance neurotransmitter production associated with pain syndromes is limited by multiple factors, specifically unavailability of adequate essential amino acids in the diet and increased turnover rates of amino acids needed to produce neurotransmitters in pain syndromes. Other factors such as prolonged pharmaceutical use deplete the nerve cells of neurotransmitters. Attempts to modify brain neurochemistry have focused on single neurotransmitters such as serotonin or GABA. However, this approach fails to address the complexity and complementary influences of multiple neurotransmitters on patient perception of pain and suffering.

Theramine is a proprietary prescription Medical Food which concurrently enhances several neurotransmitters that are involved in pain modulation and sensation by providing neurotransmitter precursors in the form of amino acids, (see attached Monograph for detailed discussion). Small trials have found Theramine effective in reducing and modifying pain without demonstrable side effects. Theramine simultaneously stimulates the production of the neurotransmitters serotonin, GABA, brain induced cortisol, nitric oxide, and glutamate.

ELIGIBILITY:
Inclusion Criteria:

1. Back pain lasting greater than six (6) weeks. Pain must be present on at least 5 out of 7 days during each of the two weeks prior to screening visit
2. Analgesic medication used to treat pain at least 4 out of last 7 days and at least 10 days in the last month
3. Men and non-pregnant, non-lactating women over the age of 18 and under the age of 75, able to read, understand and sign English-language informed consent, with diagnosis of back pain and baseline back pain greater than 40 mm out of 100 mm on visual analog scale
4. Those taking an NSAID for pain must discontinue use during a washout period based on the attached five (5) half-lives of drug chart
5. If undergoing physical therapy for back pain, therapy must be stable at least three (3) weeks prior to study and remain the same throughout study
6. If using psychoactive medication which might have analgesic effects, (i.e. anti-depressants or anti-convulsants-), treatment must be stable for at least three (3) months prior to study
7. For men and women of child-bearing potential, must be willing to use adequate contraception and not be pregnant or impregnate their partner during the entire time of study
8. Must be willing to commit to all clinical visits during study-related procedures, including required discontinuation (washout) of analgesic or anti-inflammatory medication prior to Day 1 randomization. The patient must agree to using acetaminophen for rescue medication

Exclusion Criteria:

1. Patients with back surgery in the past six (6) months
2. Patients with significant neurologic impairment, as diagnosed on screening physical examination
3. Patients with evidence or history of fracture of the spine in the past year
4. Patients not fluent in English
5. Use of aspirin for non-arthritic conditions, unless at a dose less than or equal to 325 mg a day, and must be stable for at least one (1) month prior to screening
6. Use of controlled substances and/or opiate analgesic for pain, for more than 5 days within the last 30 days prior to screening visit
7. Receipt of an oral intramuscular or soft-tissue injection of corticosteroid within one (1) month prior to screening
8. Participation in a clinical trial within the one (1) month prior to screening
9. History of epidurals in the past three (3) months
10. History of alcohol or substance abuse
11. Uncontrolled or unstable serious cardiovascular, pulmonary, gastrointestinal or urogenital, endocrine, neurologic or psychiatric disorder
12. History of gastrointestinal bleed or documented gastric or duodenal ulcer

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2010-09; Primary Completion 2011-02 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Roland-Morris Lower Back Pain Scale | 28 Days
  The primary efficacy outcome will be the change from baseline in awakening stiffness and pain subscale scores obtained from the Roland-Morris Lower Back Pain.

SECONDARY OUTCOMES:
Visual Analog Scale Evaluation | 28 days
  The primary efficacy outcome will be the change from baseline in awakening stiffness and pain subscale scores obtained from the Visual Analog Scale Evaluation.
Oswestry Low Back Pain Scale | 28 Days
  Functionality outcomes obtained from the Oswestry Low Back Pain Scale
C-reactive protein | 28 Days
  Percent change in c-reactive protein levels from baseline to Day 28.
Interleukin-6 | 28 Days
  Percent change in Il-6 level from baseline to Day 28.
Amino Acid Panel | 28 Days
  Change in amino acid turnover rate from baseline to Day 28.

CONTACTS AND LOCATIONS:
Locations (1):
- Targeted Medical Pharma, Los Angeles, California, United States

REFERENCES:
- See also: Targeted Medical Pharma — http://tmedpharma.com